CLINICAL TRIAL: NCT01866111
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Dose-Response Trial of YKP3089 as Adjunctive Therapy in Subjects With Partial Onset Seizures, With Optional Open-Label Extension
Brief Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 2 Trial of YKP3089 as Adjunctive Therapy in Subjects With Partial Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP3089C017
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2022-04-29 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Cenobamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- YKP3089 Low Dose (Experimental): YKP3089 Low Dose
  Interventions: Drug: YKP3089
- YKP3089 Medium Dose (Experimental): YKP3089 Medium Dose
  Interventions: Drug: YKP3089
- YKP3089 High Dose (Experimental): YKP3089 High Dose
  Interventions: Drug: YKP3089

INTERVENTIONS:
Drug: YKP3089
  Arms: YKP3089 High Dose; YKP3089 Low Dose; YKP3089 Medium Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled dose response study, with an 8-week prospective baseline and an 18 week double-blind treatment period (including a 6-week titration phase and 12 week maintenance phase), followed by a 3-week blinded study drug taper period (for subjects leaving the study) or a 2-week blinded conversion period (for subjects who will participate in the open-label extension).

The primary objective of this study is to determine the effective dose range of YKP3089 as adjunctive therapy for the treatment of partial seizures.

The trial will also evaluate the safety and tolerability of YKP3089 in the partial epilepsy population.

ELIGIBILITY:
Inclusion Criteria:

* Weight at least 40 kg
* A diagnosis of partial epilepsy according to the International League Against Epilepsy's Classification of Epileptic Seizures. Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history)
* Have uncontrolled partial seizures despite having been treated with at least 1 AED within approximately the last 2 years
* During the 8-week baseline period, subjects must have at least 8 partial seizures including only simple partial seizures with motor component, complex partial seizures, or secondarily generalized seizures without a seizure-free interval of greater than 25 days any time during the 8 weeks baseline. Subjects must have at least 3 of these partial seizures during each of the two consecutive 4-week segments of the baseline period
* Currently on stable antiepileptic treatment regimen.

Exclusion Criteria:

* A history of nonepileptic or psychogenic seizures
* Presence of only nonmotor simple partial seizures or primary generalized epilepsies
* Presence or previous history of Lennox-Gastaut syndrome
* An active CNS infection, demyelinating disease, degenerative neurologic disease, or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
* Any clinically significant psychiatric illness, psychological, or behavioral problems that, in the opinion of the Investigator, would interfere with the subject's ability to participate in the study
* History of alcoholism, drug abuse, or drug addiction within the past 2 years
* History of status epilepticus within 3 months of Visit 1
* A "yes" answer to Question 1 or 2 of the C-SSRS (Baseline/Screening version) Ideation Section in the past 6 months or a "yes" answer to any of the Suicidal Behavior Questions in the past 2 years
* More than 1 lifetime suicide attempt
* Participation in any other trials involving an investigational product or device within 30 days of screening (or longer, as required by local regulations)
* A history of any previous exposure to YKP3089

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (21):
  - St. Joseph's Hospital and Medical Center - Barrow Neurology Clinics, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Kaiser Permanente, Department of Neurology, Anaheim, California
  - Neuro-Pain Medical Center, Fresno, California
  - West Los Angeles VA Medical Center, Clinical Research Center, Los Angeles, California
  - Neuroresearch, Inc. - Torrance, Torrance, California
  - Neuroresearch II, Inc., Ventura, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Lovelace Scientific Resources, Inc., Sarasota, Florida
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Johns Hopkins University, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Neurology Clinic PC, Waldorf, Maryland
  - The Comprehensive Epilepsy Care Center for Children and Adults, St Louis, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - NYU Comprehensive Epilepsy Center, New York, New York
  - The Neurological Institute, PA, Charlotte, North Carolina
  - Thomas Jefferson Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Vanderbilt Epilepsy Clinic, Nashville, Tennessee
  - Austin Epilepsy Care Center, Austin, Texas
  - University of Virginia Comprehensive Epilepsy Program, Charlottesville, Virginia
- Australia (5):
  - Institute of Neurological Sciences, Prince of Wales Hospital, Randwick, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Epilepsy Research Centre, Melbourne Brain Centre, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Bulgaria (3):
  - University Multiprofile Hpspital for Active Treatment "Sveti Georgi" EAD, Clinic of Neurological Diseases, Plovdiv
  - "First Multiprofile Hospital for Active Treatment - Sofia" EAD, Neurology Clinic, Sofia
  - University of Multiprofile Hospital for Active Treatment "Aleksandrovska" EAD, Clinic of Neurological Diseases, Sofia
- Czechia (3):
  - Fakultní nemocnice Ostrava, Neurologická klinika, Ostrava
  - Mediscan Group, s.r.o, Prague
  - Fakultni nemocnice v Motole, Neurologická klinika, Prague
- France (2):
  - CHU - Service Neurophysiologie Clinique, Dijon
  - Hôpital Central - CHU de Nancy - Service de Neurologie, Nancy
- Germany (3):
  - Epilepsiezentrum Berlin- Bradenburg, Epilepsieklinik "Tabor", Bernau bei Berlin
  - Krankenhaus Mara gGmbH, Epilepsiezentrum Bethel, Bielefeld
  - Epilepsiezentrum Kork, Kehl
- Országos Klinikai Idegtudományi Intézet, Budapest, Hungary
- Israel (3):
  - Department of Neurology, Hadassah University Hospital Ein Kerem, Kiryat Hadassah, Jerusalem
  - Western Galilee Hospital, Department of Neurology, Nahariya
  - The Chaim Sheba Medical Center, Department of Neurology, Ramat Gan
- Poland (5):
  - M.A. - LEK A.M. Maciejowscy S.C. Centrum Terapii SM, Katowice
  - NOVO-MED Zielinski I Wspolnicy Spolka Jawna, Katowice
  - NZOZ Centrum Medyczne "Dendryt", Katowice
  - Fundacja Epileptologii profesora Jerzego Majkowskiego, Warsaw
  - Instytut Psychaitrii I Neurologii, II Klinika Neurologiczna, Warsaw
- Romania (2):
  - Roceanu Adina Maria Neurology Individual Medical Center, Bucharest
  - Sapiens Medical Center SRL, Bucharest
- Serbia (3):
  - Clinical of Neurology, Clinical Center of Serbia, Belgrade
  - Institute of Mental Health, Belgrade
  - Clinical Hospital Center Kragujevac, Kragujevac
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (5):
  - Hospital Universitario San Cecilio - Servicio de Neurologia, Granada
  - Hospital Ruber Internacional - Programa Epilepsia, Madrid
  - Fundación Jiminez Diaz-Servicio de Neurologia, Madrid
  - Hospital Clinico Universitario San Carlos, Serv. Neurologia, Madrid
  - Hospital Universitario y Politecnico La Fe - Servicio Neurologia, Valencia
- Srinagarind Hospital, Na Muang, Changwat Khon Kaen, Thailand
- Ukraine (5):
  - Neurology of Kharkiv Medical Academy of Postgraduate Education based on Department of Neurology #3 of State Treatment and Prevention Institution "Central Clinical Hospital of Ukrzaliznytsya", Kharkiv
  - TDC "Epilepsy" based on Department #19 of Kiev Territorial Medical Association "Psychiatry", Kyiv
  - Lviv Regional Antiepileptic Center based on Department of Neurology of Lviv Regional Clinical Hospital and Chair of Neurology of Lviv National Medical University n.a. Danylo Galytskyy, Lviv
  - MI "Odessa Regional Clinical Hospital," Neurological and Neurosurgical Center based on Neurosurgery Department, Odesa
  - Department #2 of Regional Clinical Center of Neurosurgery and Neurology, Uzhhorod

REFERENCES:
- [Derived] Klein P, Aboumatar S, Brandt C, Dong F, Krauss GL, Mizne S, Sanchez-Alvarez JC, Steinhoff BJ, Villanueva V. Long-term Efficacy and Safety From an Open-Label Extension of Adjunctive Cenobamate in Patients With Uncontrolled Focal Seizures. Neurology. 2022 Sep 5;99(10):e989-e998. doi: 10.1212/WNL.0000000000200792. PMID 35705501
- [Derived] Rosenfeld WE, Nisman A, Ferrari L. Efficacy of adjunctive cenobamate based on number of concomitant antiseizure medications, seizure frequency, and epilepsy duration at baseline: A post-hoc analysis of a randomized clinical study. Epilepsy Res. 2021 May;172:106592. doi: 10.1016/j.eplepsyres.2021.106592. Epub 2021 Feb 18. PMID 33662894
- [Derived] Krauss GL, Klein P, Brandt C, Lee SK, Milanov I, Milovanovic M, Steinhoff BJ, Kamin M. Safety and efficacy of adjunctive cenobamate (YKP3089) in patients with uncontrolled focal seizures: a multicentre, double-blind, randomised, placebo-controlled, dose-response trial. Lancet Neurol. 2020 Jan;19(1):38-48. doi: 10.1016/S1474-4422(19)30399-0. Epub 2019 Nov 14. PMID 31734103
- [Derived] Bialer M, Johannessen SI, Levy RH, Perucca E, Tomson T, White HS. Progress report on new antiepileptic drugs: A summary of the Twelfth Eilat Conference (EILAT XII). Epilepsy Res. 2015 Mar;111:85-141. doi: 10.1016/j.eplepsyres.2015.01.001. Epub 2015 Jan 19. PMID 25769377

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 533 subjects were screened and 96 were excluded for the following reasons: did not meet eligibility criteria (n=83) and withdrew consent (n=13).
Groups:
- Placebo: Subjects treated with identical appearing study drug.
- Cenobamate 100 mg/Day: Subjects titrated to a target dose of 100 mg/day
- Cenobamate 200 mg/Day: Subjects titrated to a target dose of 200 mg/day
- Cenobamate 400 mg/Day: Subjects titrated to a target dose of 400 mg/day
Period: Double-blind Period of Study YKP3089C017
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day
Started | 108 | 108 | 110 | 111
Completed | 94 | 95 | 90 | 81
Not Completed | 14 | 13 | 20 | 30
Not completed — Adverse Event | 5 | 12 | 15 | 23
Not completed — Withdrawal by Subject | 5 | 0 | 4 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0
Not completed — Reason Unknown | 3 | 0 | 0 | 1
Period: Open-label Extension Study YKP3089C017
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day
Started | 91 (Not all patients from Double-Blind Period consented to Open-Label Extension Period.) | 95 | 90 | 80 (Not all patients from Double-Blind Period consented to Open-Label Extension Period.)
Completed | 16 | 21 | 19 | 14
Not Completed | 75 | 74 | 71 | 66
Not completed — Adverse Event | 9 | 6 | 6 | 7
Not completed — Withdrawal by Subject | 16 | 7 | 9 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 1 | 3
Not completed — Death | 1 | 1 | 3 | 2
Not completed — Entered Expanded Access Program | 30 | 39 | 28 | 32
Not completed — Lack of Efficacy | 13 | 17 | 23 | 14
Not completed — Reason Unknown | 3 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants includes all randomized pts, 437. Baseline analysis population includes all randomized pts who took at least 1 dose of study drug with any post-baseline seizure data (434): Pbo (n=106), Cnb: 100mg (n=108), 200mg (n=109), 400mg (n=111). Baseline seizure frequency and enrollment region used analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day | Total
Number analyzed (Participants) | 108 | 108 | 110 | 111 | 437
Age, Continuous [Median (Full Range); unit: Years] | 38 [19 to 70] | 37.5 [19 to 66] | 40.5 [19 to 69] | 38.0 [21 to 66] | 38 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 56 | 59 | 216
  Male | 58 | 57 | 54 | 52 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 7 | 13 | 37
  Not Hispanic or Latino | 99 | 100 | 103 | 98 | 400
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 10 | 11 | 11 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 3 | 1 | 12
  White | 93 | 89 | 94 | 96 | 372
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 2 | 3 | 12
28-day partial-onset seizure frequency [Median (Full Range); unit: seizures/28 days] — Baseline measures were reported in the randomized population, with the exception of baseline seizure frequency/28 days, which was reported for all randomized subjects who took at least one dose of study drug and had any post-baseline seizure data. Population: Baseline seizure frequency was analyzed
  seizures/28 days
    number analyzed (Participants) | 106 | 108 | 109 | 111 | 434
    (all) | 8.4 [4 to 704] | 9.5 [3.5 to 202] | 11.0 [4 to 418] | 9.0 [4 to 638] | 9.4 [3.5 to 704]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Partial-onset Seizure Frequency Per 28 Days
Description: Percent change in complex partial and/or secondarily generalized and/or simple partial motor seizure frequency per 28 days (average 28-day seizure rate) in each treatment group during the double-blind period relative to the pretreatment baseline.
Time Frame: baseline and 18 weeks
Population: All randomly assigned patients who took at least one dose of study drug and had any post-baseline seizure data.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day
Number analyzed (Participants) | 106 | 108 | 109 | 111
percent change | -24.0 [-91 to 198] | -35.5 [-100 to 206] | -55.0 [-100 to 191] | -55.0 [-100 to 167]
Statistical Analysis 1: Comparison: Placebo vs Cenobamate 200 mg/Day; A step down procedure was used for the primary efficacy analyses to ensure the type one error rate for multiple comparisons was controlled at the 5% level using the following hierarchy: 200 mg vs placebo, 400 mg vs placebo, 100 mg vs placebo, in which a statistically significant difference had to be detected in this order for each subsequent comparison to occur; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Cenobamate 400 mg/Day; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs Cenobamate 100 mg/Day; Test type: Superiority; p = 0.007, ANCOVA

2. Secondary Outcome: 50% Responder Rate
Description: Percentage of patients achieving a 50% or more reduction from baseline in partial seizure frequency during the double-blind treatment period
Time Frame: 18 weeks
Population: All randomly assigned patients who had taken at least one dose of study drug and had any post-baseline seizure data
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day
Number analyzed (Participants) | 106 | 108 | 109 | 111
Participants | 23 | 44 | 63 | 67
Statistical Analysis 1: Comparison: Placebo vs Cenobamate 200 mg/Day; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Cenobamate 400 mg/Day; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Cenobamate 100 mg/Day; Test type: Superiority; p = 0.003, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6.75 years
Description: Adverse events were collected for each subject for 18 weeks in the double-blind period, followed by a 2-week double-blind conversion period at the beginning of the open-label extension (OLE) phase for subjects that consented to the OLE. In addition, adverse events were collected for the full duration of the OLE, with a maximum drug exposure of 331 weeks. Adverse events and serious adverse events reported below are consistent of treatment-emergent events, unless otherwise stated.
Groups:
- 100mg/Day Open-Label Extension: Subjects that consented to Open-Label Extension period of study. This includes subjects that began with a 100mg/day dose, with a target dose of 300 mg/day.
- 200mg/Day Open-Label Extension: Subjects that consented to Open-Label Extension period of study. This includes subjects that began with a 200mg/day dose, with a target dose of 300 mg/day.
- 400mg/Day Open-Label Extension: Subjects that consented to Open-Label Extension period of study. This includes subjects that began with a 400mg/day dose, with a target dose of 300 mg/day.
- Placebo Open-Label Extension: Subjects that consented to Open-Label Extension period of study. This includes subjects that began with a placebo dose, with a target dose of 300 mg/day.
Arm/Group | Placebo | Cenobamate 100 mg/Day | Cenobamate 200 mg/Day | Cenobamate 400 mg/Day | 100mg/Day Open-Label Extension | 200mg/Day Open-Label Extension | 400mg/Day Open-Label Extension | Placebo Open-Label Extension
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/108 | 0/110 | 0/111 | 1/95 | 3/90 | 3/80 | 2/91
Serious Adverse Events (participants affected / at risk) | 6/108 | 10/108 | 4/110 | 8/111 | 21/95 | 17/90 | 21/80 | 20/91
Other Adverse Events (participants affected / at risk) | 76/108 | 70/108 | 84/110 | 100/111 | 87/95 | 80/90 | 70/70 | 80/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Cenobamate 100 mg/Day (N=108) | Cenobamate 200 mg/Day (N=110) | Cenobamate 400 mg/Day (N=111) | 100mg/Day Open-Label Extension (N=95) | 200mg/Day Open-Label Extension (N=90) | 400mg/Day Open-Label Extension (N=80) | Placebo Open-Label Extension (N=91)
Seizure (Nervous system disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 2 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ALT increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
AST increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DRESS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Entercolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden unexplained death in epilepsy (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cranicerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Seizure cluster (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebellar haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postictal headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychogenic seizure (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Psychomotor retardation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — Non-treatment emergent AE.
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — Non-treatment emergent AE.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=108) | Cenobamate 100 mg/Day (N=108) | Cenobamate 200 mg/Day (N=110) | Cenobamate 400 mg/Day (N=111) | 100mg/Day Open-Label Extension (N=95) | 200mg/Day Open-Label Extension (N=90) | 400mg/Day Open-Label Extension (N=70) | Placebo Open-Label Extension (N=80)
Somnolence (Nervous system disorders) | 9 | 20 | 23 | 41 | 24 | 29 | 26 | 32
Dizziness (Nervous system disorders) | 15 | 19 | 22 | 37 | 43 | 29 | 26 | 30
Headache (Nervous system disorders) | 6 | 11 | 12 | 12 | 21 | 16 | 9 | 13
Balance disorder (Nervous system disorders) | 0 | 3 | 2 | 10 | 7 | 4 | 3 | 7
Nystagmus (Nervous system disorders) | 1 | 3 | 4 | 7 | 7 | 4 | 3 | 9
Ataxia (Nervous system disorders) | 1 | 2 | 4 | 7 | 7 | 4 | 1 | 7
Dysarthria (Nervous system disorders) | 0 | 2 | 3 | 7 | 6 | 5 | 3 | 5
Fatigue (General disorders) | 9 | 13 | 19 | 27 | 18 | 18 | 8 | 15
Gait disturbance (General disorders) | 3 | 1 | 6 | 9 | 15 | 8 | 12 | 10
Diplopia (Eye disorders) | 2 | 8 | 11 | 17 | 17 | 12 | 9 | 14
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 10 | 7 | 5 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 7 | 1 | 10 | 7 | 5 | 4 | 8
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 6 | 12 | 3 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 4 | 4 | 11 | 5 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 4 | 3 | 11 | 11 | 8 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 6 | 9 | 7 | 6 | 4
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 3 | 6 | 7 | 5 | 5 | 13
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 6 | 3 | 5 | 5 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 5 | 1 | 6 | 5
Nasopharyngitis (Infections and infestations) | 5 | 2 | 2 | 5 | 11 | 6 | 10 | 5
Laceration (Injury, poisoning and procedural complications) | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 2 | 2 | 2 | 1 | 8 | 2 | 8 | 7
Memory impairment (Nervous system disorders) | 1 | 2 | 3 | 2 | 8 | 5 | 2 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 5 | 4 | 4 | 4
Urinary tract infection (Infections and infestations) | 1 | 2 | 3 | 0 | 4 | 7 | 5 | 8
Sinusitis (Infections and infestations) | 2 | 0 | 2 | 1 | 3 | 3 | 0 | 6
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 0 | 2 | 7
Influenza (Infections and infestations) | 4 | 1 | 3 | 0 | 4 | 2 | 0 | 5
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 4 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 3 | 3 | 6 | 4 | 4 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 5
Insomnia (Psychiatric disorders) | 2 | 0 | 3 | 1 | 1 | 7 | 2 | 4
Confusional state (Psychiatric disorders) | 0 | 2 | 2 | 3 | 2 | 1 | 4 | 0
Vision blurred (Eye disorders) | 0 | 2 | 2 | 4 | 5 | 5 | 1 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 5 | 4 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 5 | 0 | 4 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 2 | 5 | 1 | 2 | 1
Weight decreased (Investigations) | 0 | 2 | 0 | 1 | 7 | 3 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 3 | 2 | 5
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT01866111/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT01866111/SAP_001.pdf